CLINICAL TRIAL: NCT02405403
Title: Microglial Activation Role In ALS (MARIA)
Acronym: MARIA
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: It was more difficult than planned to find patients filling inclusion criteria and those which corresponded didn't agree to participate
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PHAO-13-PC/MARIA
Record Dates: First submitted 2015-03-02; First posted 2015-04-01 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis disease; PET; microglial activation
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- amyotrophic lateral sclerosis (ALS) (Experimental): [18F]DPA-714 PET
  Interventions: Drug: [18F]DPA-714 PET

INTERVENTIONS:
Drug: [18F]DPA-714 PET — [18F]DPA-714 Positron Emission Tomography
  Other Names: [18F]DPA-714

SUMMARY:
Neuroinflammation, characterized in particular by microglia activation, is an essential component of Amyotrophic Lateral Sclerosis (ALS) pathogenesis. Translocator Protein (TSPO) is recognized as a specific and sensitive biomarker of neuroinflammation, reflecting disease activity. An experimental radiopharmaceutical specific of TSPO expression, namely [18F]DPA714, allow to quantify this microglial activation using Positon Emission Tomography (PET) imaging.

The purpose of this study is to longitudinally correlate the spatial distribution of neuroinflammation with the pro- or anti-inflammatory state of activated microglia cells in ALS, in order to evaluate neurotoxic or neuroprotective microglia activity, by complementary approaches in 20 ALS patients:

* in vitro: measuring concentrations of several pro- and anti-inflammatory cytokines secreted by microglial cells in the cerebrospinal fluid (CSF).
* in vivo: [18F]DPA714 PET imaging. These assays will be performed in the framework of the clinical follow-up of ALS patients, at the diagnosis of ALS disease and 6 months latter.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥ 18 years old
* Patient with probable or definite sporadic Amyotrophic Lateral Sclerosis (ALS) form according to the modified criteria of El Escorial
* Treated with riluzole 2 weeks
* Evolution less than 18 months
* Mini-Mental State Examination (MMS) score ≥ 26 and Frontal Assessment Battery (FAB) (normal)
* Affiliated to a social security system

Exclusion Criteria:

* Another unbalanced progressive pathology
* Vascular diseases (hypertension, diabetes, smoking, dyslipidemia) unbalanced
* Forced vital capacity <75%
* Weight loss> 10% of the weight before disease
* Status "low affinity binder" or "mixed affinity binder", the TSPO respect to the [18 F] DPA-714, which can interfere with the process of neuroinflammation: drugs with anti-inflammatory drugs (NSAIDs, corticosteroids, azathioprine, anti-tumor necrosis factor (TNF), antibiotics)
* Benzodiazepine in the week before the PET scan [18F] DPA-714 given the potential consequences for TSPO receivers
* Contraindications to MRI in patients with:

  1. Metallic foreign body eye.
  2. Any implanted electronic medical irremovably (pacemaker, neurostimulator, cochlear implants ...)
  3. Metal heart valve,
  4. Vascular clips formerly located on cranial aneurysm.
* Treatment in the month before the PET scan [18F] DPA-714 antagonist N-methyl-D-aspartate (NMDA) (memantine)
* Pregnant women, lactating women, and women in age for procreation and without reliable contraception or without history of hysterectomy
* ◦Person under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03 (Estimated); Primary Completion 2016-09 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Concentration of cytokines in cerebrospinal fluid (pg/mL) | 18 months

SECONDARY OUTCOMES:
Fixation and distribution of [18F]DPA-714 (Binding Potential BP) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CORCIA, PhD, Principal Investigator — CHRU TOURS
Locations (1):
- University Hospital, Tours, France

REFERENCES:
- [Result] Corcia P, Valdmanis P, Millecamps S, Lionnet C, Blasco H, Mouzat K, Daoud H, Belzil V, Morales R, Pageot N, Danel-Brunaud V, Vandenberghe N, Pradat PF, Couratier P, Salachas F, Lumbroso S, Rouleau GA, Meininger V, Camu W. Phenotype and genotype analysis in amyotrophic lateral sclerosis with TARDBP gene mutations. Neurology. 2012 May 8;78(19):1519-26. doi: 10.1212/WNL.0b013e3182553c88. Epub 2012 Apr 25. PMID 22539580
- [Result] Blasco H, Corcia P, Moreau C, Veau S, Fournier C, Vourc'h P, Emond P, Gordon P, Pradat PF, Praline J, Devos D, Nadal-Desbarats L, Andres CR. 1H-NMR-based metabolomic profiling of CSF in early amyotrophic lateral sclerosis. PLoS One. 2010 Oct 8;5(10):e13223. doi: 10.1371/journal.pone.0013223. PMID 20949041
- [Result] Arlicot N, Vercouillie J, Ribeiro MJ, Tauber C, Venel Y, Baulieu JL, Maia S, Corcia P, Stabin MG, Reynolds A, Kassiou M, Guilloteau D. Initial evaluation in healthy humans of [18F]DPA-714, a potential PET biomarker for neuroinflammation. Nucl Med Biol. 2012 May;39(4):570-8. doi: 10.1016/j.nucmedbio.2011.10.012. Epub 2011 Dec 14. PMID 22172392
- [Result] Corcia P, Ingre C, Blasco H, Press R, Praline J, Antar C, Veyrat-Durebex C, Guettard YO, Camu W, Andersen PM, Vourc'h P, Andres CR. Homozygous SMN2 deletion is a protective factor in the Swedish ALS population. Eur J Hum Genet. 2012 May;20(5):588-91. doi: 10.1038/ejhg.2011.255. Epub 2012 Jan 25. PMID 22274580
- [Result] Corcia P, Tauber C, Vercoullie J, Arlicot N, Prunier C, Praline J, Nicolas G, Venel Y, Hommet C, Baulieu JL, Cottier JP, Roussel C, Kassiou M, Guilloteau D, Ribeiro MJ. Molecular imaging of microglial activation in amyotrophic lateral sclerosis. PLoS One. 2012;7(12):e52941. doi: 10.1371/journal.pone.0052941. Epub 2012 Dec 31. PMID 23300829